CLINICAL TRIAL: NCT00693628
Title: Effects of Shrinker Use on Healing and Volume for Transtibial Amputees
Brief Title: Effects of Shrinker Use on Healing and Volume
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of enrollment
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13310; 13310 (Other: University of Oklahoma Health Sciences Center)
Record Dates: First submitted 2007-12-20; First posted 2008-06-09 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Transtibial Amputation
Keywords: volume; healing; shrinker; transtibial amputation; individuals who have undergone transtibial amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shrinker (Active Comparator): Patients receive 20-30 mmHg compression shrinker, an elastic compression garment that is worn on the residual limb and is used to reduce edema and promote healing.
  Interventions: Device: compression shrinker
- No Shrinker (No Intervention): Control group - participants will not receive an intervention (compression shrinker).
- Shrinker 2 (Active Comparator): Patients receive 30-40 mmHg compression shrinker, an elastic compression garment that is worn on the residual limb and is used to reduce edema and promote healing.
  Interventions: Device: compression shrinker

INTERVENTIONS:
Device: compression shrinker — Two levels of compression: 20-30 mmHg or 30-40 mmHg shrinker
  Other Names: Juzo® Compression Therapy Garment
  Arms: Shrinker; Shrinker 2

SUMMARY:
We expect subjects in the interventional groups, who wear shrinkers, to heal more quickly than control subjects who wear no shrinkers. We also expect them to experience greater reduction in residual limb volume during the early stages of postoperative care leading up to prosthetic fitting, fewer healing complications, reduced time to the prosthetic fitting, increased time to the first prosthetic socket replacement, and fewer socket replacements by the end of the "transition to stable phase".

DETAILED DESCRIPTION:
Edema is an inevitable result of amputation surgery. Persistent edema can affect oxygen and nutrient flow into, as well as waste flow out of the residual limb. Shrinkers are a common and effective treatment for edema. However, their influence on healing and long term limb volume has not been studied. This study will pertain to human subjects affected by primary transtibial amputation. Two interventional groups of patients will use shrinkers with different levels of compression as part of their rehabilitation. A third, control group will not use shrinkers. The groups will be studied to determine the effects of shrinker use on healing and long term residual limb volume.

ELIGIBILITY:
Inclusion Criteria:

* Recently undergone primary transtibial amputation
* Patients between ages of 18 and 100 years of age

Exclusion Criteria:

* Undergone previous amputations above the Symes level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Day, BSPO, Principal Investigator — University of Oklahoma Health Sciences Center Department of Orthopedic Surgery & Rehabilitation, Division of Orthotics & Prosthetics
Locations (1):
- University of Oklahoma Health Sciences Center, O'Donoghue Orthotics & Prosthetics Clinic, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Shrinker: Patients receive 20-30 mmHg or 30-40 mmHg shrinker, an elastic compression garment that is worn on the residual limb and is used to reduce edema and promote healing.
  compression shrinker: Two levels of compression: 20-30 mmHg or 30-40 mmHg shrinker
- No Shrinker: Patients will receive no shrinker
Period: Overall Study
Arm/Group | Shrinker | No Shrinker
Started | 0 (No data is available indicating to which group patients were assigned.) | 0 (No data is available indicating to which group patients were assigned .)
Completed | 0 (Only 4 patients enrolled in study. No data indicating their group assignment) | 0 (Only 4 patients enrolled in study. No data indicating their group assignment.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Early termination of the study due to poor enrollment numbers, i.e., only 4 subjects were enrolled. No analysis was performed due to insufficient data to assess outcome measures. The number of patients in each group is unknown.
Groups:
- Total: Total of all reporting groups
Arm/Group | Shrinker | No Shrinker | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
  <=18 years |  |  | 0
  Between 18 and 65 years |  |  | 0
  >=65 years |  |  | 0
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Time to Healing
Description: time to healing in each group
Time Frame: 1 year
Population: study was closed due to low enrollment. Data were not collected.
Arm/Group | Shrinker | No Shrinker
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed due to early termination.
Arm/Group | Shrinker | No Shrinker
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination of the study due to poor enrollment numbers, (only 4 subjects were enrolled). No analysis was performed due to insufficient data to assess outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes